CLINICAL TRIAL: NCT02239003
Title: NMDA-enhancing Agent for the Treatment of Mild Cognitive Impairment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chieh-Hsin Lin, Dr, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 103-3642C
Record Dates: First submitted 2014-09-09; First posted 2014-09-12 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- DAOIB (Experimental): 250-1500 mg/day, oral, for 24 weeks
  Interventions: Drug: DAOIB
- Placebo (Placebo Comparator): placebo, oral, for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DAOIB
  Arms: DAOIB
Drug: Placebo
  Arms: Placebo

SUMMARY:
NMDA neurotransmission plays an important role in learning and memory. NMDA receptors were found to decrease in the frontal lobe and hippocampus of mild cognitive impairment. This study is a randomized, double-blind, placebo-controlled drug trial. All subjects will be allocated randomly to 2 groups: (1) NMDA-enhancer: DAOIB group (starting dose: 250-500 mg/d); (2) placebo group. The study period is 24 weeks. The investigators hypothesize that DAOIB may yield better efficacy than placebo for cognitive function in patients with mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild cognitive impairment
* MMSE between 17-26
* CDR 0.5

Exclusion Criteria:

* Hachinski Ischemic Score > 4
* Substance abuse/dependence
* Parkinson disease, epilepsy, dementia with psychotic features
* Major depressive disorder
* Major physical illnesses
* Severe visual or hearing impairment

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-01; Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Alzheimer's disease assessment scale - cognitive subscale at week 8, 16 and 24 | week 0, 8, 16, 24

SECONDARY OUTCOMES:
Change from baseline in speed of processing (Category Fluency) at week 24 | week 0, 24
Change from baseline in Clinician's Interview-Based Impression of Change plus Caregiver Input at week 8, 16 and 24 | week 8, 16, 24
Change from baseline in working memory (Wechsler Memory Scale, Spatial Span) at week 24 | week 0, 24
Change from baseline in verbal learning and memory tests (Wechsler Memory Scale, Word Listing) at week 24 | week 0, 24

CONTACTS AND LOCATIONS:
Overall Officials: Chieh-Hsin Lin, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital; Hsien-Yuan Lane, MD, PhD, Study Chair — China Medical University, China
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan